CLINICAL TRIAL: NCT05824065
Title: Phase III, National, Multicenter, Randomized, Double-Blind, Superiority Clinical Trial to Evaluate the Efficacy and Safety of OMA102 in the Treatment of Female Pattern Hair Loss
Brief Title: Efficacy and Safety of OMA102 in the Treatment of Female Pattern Hair Loss
Acronym: GENERA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OMA102-III-0123
Record Dates: First submitted 2023-04-11; First posted 2023-04-21 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2023-04

CONDITIONS: Female Pattern Baldness
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OMA102 1 mg (Experimental): Ingestion of 1 oral tablet, once a day, immediately before lying down to sleep
  Interventions: Drug: OMA102
- OMA102 2 mg (Experimental): Ingestion of 1 oral tablet, once a day, immediately before lying down to sleep
  Interventions: Drug: OMA102
- Placebo (Placebo Comparator): Ingestion of 1 oral tablet, once a day, immediately before lying down to sleep
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OMA102 — 1 mg
  Arms: OMA102 1 mg
Drug: OMA102 — 2 mg
  Arms: OMA102 2 mg
Drug: Placebo — OMA102 - Placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of OMA102 1 mg and OMA102 2 mg versus placebo in the treatment of female pattern hair loss.

ELIGIBILITY:
Inclusion Criteria:

* Ability to confirm voluntary participation and agree to all trial purposes by signing and dating the informed consent forms;
* Age greater than 18 and equal or under 50 years;
* Confirmed diagnosis of female pattern hair loss, grade II to IV in Sinclair Scale;
* Participants that are disposed to maintain the same hair color, style, approximate hair length throughout the Clinical Study.

Exclusion Criteria:

* Any clinical or physical finding interpreted by the investigator as a risk to subject participation in the Clinical Study
* History of alcohol or illicit drugs abuse in the last year;
* Pregnant or breastfeeding women, who are planning to become pregnant or participants who have childbearing potential and are not using any reliable contraceptive method;
* Allergy or sensibility to any knowing components of the formula;
* Diagnosis of arterial hypertension;
* History of vasovagal syncope;
* Baseline systolic blood pressure lower than 90 mmHg and/or diastolic lower than 60 mmHg;
* Diagnosis of orthostatic hypotension (reduction of systolic blood pressure equal or superior to 20 mmHg and/or diastolic equal or superior to 10 mmHg after 3 minutes in orthostatic position);
* Body mass index (BMI) > 30 kg/m²;
* Subjects that initiated any kind of continue use medication, including contraceptives with systemic effect, until 3 months previously the inclusion in the Clinical Study;
* History of cardiovascular, liver and renal diseases;
* History of hypothyroidism, hyperthyroidism or pheochromocytoma;
* Signs or symptoms of cardiopathy or angina;
* History of edema from any etiology;
* Participants who are using tricycle antidepressants, benzodiazepines, antipsychotics, anticholinergics, sulfonamide derivatives, beta-blockers, sympathomimetics, arginine, glucocorticoid or monoamine oxidase inhibitors;
* Use of inhibitor of 5-alpha reductase or androgenic blockers in the last 12 months;
* Dermatologic diseases of the scalp, except mild seborrheic dermatitis or diagnosis of any kind of alopecia other than female pattern hair loss;
* History of surgical treatment for hair loss or presence of shaved scalp;
* Scalp microinfusion, microneedling or intradermotherapy in the last 3 years;
* Vaginal or cesarean deliveries 6 months before the inclusion in the study;
* Drastic modification of habitual diet, as food restrictions or hyperselectivity;
* Current cancer or history of cancer in the last 5 years;
* Participation in others research protocols in the last 12 months, unless the investigator judges that there may be a direct benefit to the participant.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 504 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of OMA102 1 mg and OMA102 2 mg in the promotion of hair growth in the mid front area assessed by digital phototrichogram. | 6 months
  Variation of hair in the mid-front area after 6 months of treatment in comparison to baseline, assessed by digital phototrichogram.

SECONDARY OUTCOMES:
Efficacy of OMA102 1 mg and OMA102 2 mg in the promotion of hair growth in the mid front area assessed by digital phototrichogram. | 3 months
  Variation of hair in the mid-front area after 3 months of treatment in comparison to baseline, assessed by digital phototrichogram.
Efficacy of OMA102 1 mg and OMA102 2 mg in the promotion of non vellus and vellus hair growth, in the mid frontal area, assessed by digital phototrichogram. | 3 and 6 months
  Variation of non vellus and vellus hair in the mid-front area after 3 and 6 months of treatment in comparison to baseline, assessed by digital phototrichogram.
Efficacy of OMA102 1 mg and OMA102 2 mg in the proportion of subjects with an improvement of global photographs, assessed by Clinical Global Impression of Improvement (CGI-I) by the investigator perception. | 3 and 6 months
  Efficacy of OMA102 1 mg and OMA102 2 mg in the proportion of subjects with an improvement global photographs assessed by Clinical Global Impression of Improvement (CGI-I) by the investigator perception, 3 and 6 months after treatment.
Efficacy of OMA102 1 mg and OMA102 2 mg in the proportion of subjects with an improvement of global photographs, assessed by Patient Global Impression, PGI-I, by the subject perception. | 3 and 6 months
  Efficacy of OMA102 1 mg and OMA102 2 mg in the proportion of subjects with an improvement of Global Photographs assessed by Patient Global Impression PGI-I, by the investigator perception, 3 and 6 months after treatment.
Efficacy of OMA102 1 mg and OMA102 2 mg in quality of life, assessed by Women's Androgenetic Alopecia Quality of Life (WAA-QoL). | 3 and 6 months
  Efficacy of OMA102 1 mg and OMA102 2 mg in quality of life, assessed by Women's Androgenetic Alopecia Quality of Life (WAA-QoL) in comparison to baseline, 3 and 6 months after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- EMS, Hortolândia, São Paulo, Brazil